CLINICAL TRIAL: NCT03731416
Title: Ridge Augmentation in Atrophic Anterior Maxillary Ridges With Native Collagen Membrane and Anorganic Bovine Bone Derived Mineral With and Without Particulated Autogenous Bone Chips
Brief Title: Guided Bone Regeneration in Atrophic Anterior Maxillary Ridges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hossam samir mohamed ahmed elbaha, Principal Investigator(doctor), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Guided bone regeneration
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Bone Resorption Disorder
Keywords: GBR, autogenous bone, xenograft

STUDY DESIGN:
Intervention Model Description: The patients will be randomly divided into 2 equal groups
Who Masked: Investigator
Masking Description: Each patient will be given a code by the researcher and the observers will be blind to which group this case belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GBR by xenograft (Placebo Comparator): * Patients of both groups will be subjected to CBCT (diagnostic for upper arch).
  * Intra operative procedures (for both groups) followed by CBCT will be taken for every patient.
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  * Flap will be done.
  * In the study group: bone decortication will be done using surgical round bur, anorganic bovine bone derived mineral will be packed then covered at the defected area by a native collagen membrane which will be stabilized by tacks.
  * • The site will then be copiously irrigated with saline in preparation for closure.
  * The flap will then be closed using interrupted 4/0 resorbable sutures.
  Interventions: Procedure: GBR by xenograft and autogenous bone
- GBR by xenograft ,autogenous bone (Active Comparator): Intervention In the control group:first crestal incision then two vertical incisions by blade 15c,full thickness flap reflection, bone decortication will be done using surgical round bur, autogenous bone will be harvested by trephine bur ,mixed 1:1 with anorganic bovine bone derived mineral and packed at the defected area(atrophic maxilla) then covered by a native collagen membrane which will be stabilized by tacks.Then The flap will then be closed using interrupted 4/0 resorbable sutures.
  Interventions: Procedure: GBR by xenograft and autogenous bone

INTERVENTIONS:
Procedure: GBR by xenograft and autogenous bone — Ridge augmentation by native collagen membrane and mix of anorganic bovine bone derived mineral with particulated autogenous bone chips (ratio 1:1).

SUMMARY:
This study is aiming to evaluate clinically, radiographically ,and histologically GBR using collagen membrane in combination with a mixture of ABBM and autogenous particulated bone compared to collagen membrane with ABBM in atrophied anterior maxilla.

DETAILED DESCRIPTION:
Guided bone regeneration (GBR) has been proposed as a possible alternative for patients with severe horizontal bone atrophy, to overcome the drawback of bone blocks techniques.6,8 To protect and prevent the invasion of the clot by nonosteogenic cells, maintaining an adequate biological space for the regeneration of bone tissue, the use of resorbable membranes, in combination with autologous or heterologous particulate bone have been proposed. Expanded polytetrafluoroethylene (e-PTFE) membranes are the most used non-resorbable membranes with the longest published follow-up, considering them the gold standard in the reconstructions of major horizontal bone defects. However, a second surgery is needed to remove them and they may get exposed in the oral cavity and contaminate with possible infection and graft loss. Conversely, the resorbable membranes most advantages are an ability to merge with the host tissues, as well as a rapid resorption in case of exposure, thereby reducing the risk of bacterial contamination. Resorbable membranes in combination with particulated anorganic bovine bone (ABB) can be used for the augmentation of horizontally deficient ridges. Particulated autogenous bone can be mixed with bone substitutes to add more osteogenic factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophied anterior maxillary ridge area.
* Age: 18 years and older.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate bone augmentation

Exclusion Criteria:

* • Heavy smokers more than 20 cigarettes per day.(32)

  * Patients with systemic disease that may affect normal healing.
  * Psychiatric problems.
  * Disorders to bone augmentation are related to history of radiation therapy to the head and neck neoplasia.
  * Pregnant or nursing women.
  * Patients with uncontrolled diabetes mellitus, rheumatoid arthritis or osteoporosis.
  * Patient with previous history of radiotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-12 (Estimated)

PRIMARY OUTCOMES:
Height and width of bone gained | 6 months
  Height and width of bone gained in mm by CBCT

SECONDARY OUTCOMES:
Bone area percentage | 6 months
  Bone area percentage % by Histo-morphometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: hossam Elbaha, Study Chair — Cairo University

REFERENCES:
- [Result] Meloni SM, Jovanovic SA, Urban I, Canullo L, Pisano M, Tallarico M. Horizontal Ridge Augmentation using GBR with a Native Collagen Membrane and 1:1 Ratio of Particulated Xenograft and Autologous Bone: A 1-Year Prospective Clinical Study. Clin Implant Dent Relat Res. 2017 Feb;19(1):38-45. doi: 10.1111/cid.12429. Epub 2016 Jun 9. PMID 27283920
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pubmed/27283920